CLINICAL TRIAL: NCT07037745
Title: The Effect of Intravenous Dexamethasone in Addition to Intrathecal Morphine on Postoperative Analgesia and Nausea/Vomiting in Geriatric Hip Fractures: A Retrospective Study
Brief Title: Dexamethasone + Intrathecal Morphine in Hip Fractures
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kadir Arslan, Specialist physician, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2024.09.185
Record Dates: First submitted 2025-06-15; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-09

CONDITIONS: Hip Fracture Surgeries
Keywords: postoperative pain; hip fracture; geriatric; spinal morphine; multimodale analgesia
MeSH Terms: conditions — Pain, Postoperative; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group D: Group that received 0.1 mg intrathecal morphine and 8 mg intravenous dexamethasone
- Group C: 0.1 mg intrathecal morphine and 8 mg intravenous dexamethasone were not administered in the group, control group

SUMMARY:
Hip fractures (proximal femur fractures) are a global public health problem with high morbidity and mortality rates, especially in the geriatric population aged 65 years and older. Hip fractures, an important consequence of osteoporosis, occur as a result of low-energy trauma with advancing age. Increased mortality rates are associated with an increased risk of postoperative complications, the need for an intensive care unit, prolonged hospital stay, and decreased quality of life.

Multimodal analgesia strategies in geriatric hip fracture patients aim to provide adequate pain control while limiting systemic opioid use. Spinal anesthesia, one of the neuraxial anesthesia methods, is frequently used in this patient group, as it avoids complications associated with general anesthesia. It has been reported that the addition of intrathecal morphine (ITM) to local anesthetics used in minimal-dose spinal anesthesia is practical in postoperative pain control. It has been reported that the use of ITM in the dose range of 0.1-0.2 mg in major orthopedic surgeries such as total hip arthroplasty significantly reduces systemic opioid use and provides a decrease in early pain scores. Nausea, vomiting, and decreased gastrointestinal function in the postoperative period may impair patient comfort. In addition, depending on the dose used, ITM may cause side effects such as postoperative nausea and vomiting (PONV) and pruritus. It has been reported that perioperative use of intravenous dexamethasone reduces postoperative pain scores and the consumed analgesic dose in patients undergoing spinal anesthesia using ITM, as well as reducing PONV. Although the benefit of opioid-sparing analgesia provided by ITM in geriatric hip fracture patients is important, the role of intravenous dexamethasone in effectively controlling side effects such as nausea, vomiting, and pruritus, which may increase with it, is a current and critical area of research.

This study aimed to investigate the effect of intravenous (8 mg) dexamethasone added to intrathecal morphine (0.1 mg) on postoperative pain scores, opioid consumption, PONV, and pruritus in geriatric hip fracture patients.

DETAILED DESCRIPTION:
The study is a retrospective cohort study conducted in a tertiary center. In our clinic, hip fracture operations are frequently performed under spinal anesthesia using ITM in geriatric hip fracture patients. In this study, the effects of intravenous 8 mg dexamethasone on analgesia scores, PONV, and pruritus adverse effects in geriatric hip fracture patients under spinal anesthesia using 0.1 mg ITM will be investigated.

Pain scores, PONV, and pruritus parameters of hip fracture patients who were and were not administered intravenous 8 mg dexamethasone after spinal anesthesia using ITM will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and above,
* both genders,
* performing hip fracture surgery under spinal anesthesia using 0.1 mg intrathecal morphine

Exclusion Criteria:

* Performing another operation with a hip fracture,
* Conversion to general anesthesia after spinal anesthesia,
* Peroperative severe cardiovascular and respiratory failure,
* Systemic steroid use,
* Uncontrolled diabetes,
* Lack of cooperation that makes it difficult to assess the level of pain and -nausea/vomiting in the postoperative period, cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric (age 65 and over) patients with hip fractures
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | 2, 6, 12, and 24 hours postoperatively
  The Visual Analog Scale (VAS) will be used to determine the intensity of pain and to compare the pain felt before and after treatment (2, 6, 12, and 24 hours postoperatively.). VAS is a reliable and easily applicable test used to measure values that cannot be easily measured numerically by converting them into a numerical format. The lowest and highest definitions of the parameters to be evaluated are written on both ends of a 100 mm line. The patient is asked to mark the most appropriate value (location) between these two extreme points. When this scale is used for pain, the numbers "0" are written on one end to indicate no pain, and "10" are written on the other end to indicate the most severe pain, and this is converted into a template, numbers between 0-10 are placed on the line, and the patient is asked to choose the closest number.

SECONDARY OUTCOMES:
Paracetamol, diclofenac sodium and tramadol consumption | First 24 hours postoperatively
  In the postoperative period, if geriatric hip fracture patients followed in the ward or intensive care unit experience pain, paracetamol 1 g (Rastamol 10mg/mL vial, Haver Farma, Turkey) is administered intravenously three times. In patients who complain of pain despite taking paracetamol, diclofenac sodium (Dichloron 75 mg/3 mL, Deva Farma, Turkey) is administered intramuscularly at a dose of 75 mg, 1 to 3 times. If there is no pain relief with diclofenac, tramadol hydrochloride (Tradolex 100 mg/2mL, Menta Farma, Turkey) can be infused in 100 mL of saline.

CONTACTS AND LOCATIONS:
Overall Officials: Kadir Arslan, M.D., Principal Investigator — University of Health Sciences Turkey, Istanbul Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Istanbul Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
No decision has been made yet. Of course, the study data will be shared if permission is received from the responsible researcher.